CLINICAL TRIAL: NCT06490237
Title: Coding of Speech Signals in the Human Auditory Nerve - an Exploratory Study
Brief Title: Coding of Speech Signals in the Human Auditory Nerve
Acronym: NeuroSpeech
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO21089
Record Dates: First submitted 2021-08-03; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Hearing Loss
Keywords: Hearing Loss; Deafness; Hearing Disorders in noise and in silence; Ear Diseases
MeSH Terms: conditions — Hearing Loss; Deafness; Ear Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with no hearing loss (Active Comparator)
  Interventions: Procedure: near field recording of human auditory nerve activity during retro sigmoid approach with contact electrode
- subjects with hearing loss (Experimental)
  Interventions: Procedure: near field recording of human auditory nerve activity during retro sigmoid approach with contact electrode

INTERVENTIONS:
Procedure: near field recording of human auditory nerve activity during retro sigmoid approach with contact electrode — During surgery using a retro-sigmoid approach in the cerebellopontine angle (microvascular decompression, vestibular neurotomy, meningioma or schwannoma removal), near-field recording of human auditory nerve activity using a contact electrode is performed on patients with normal or impaired hearing threshold.
  Each patient is explored preoperatively by hearing tests in noise and in silence. During the operation, stimuli are delivered in silence and in noise, under the same conditions as during the preoperative auditory exploration.

SUMMARY:
The fine evaluation of the function of auditory neurons in silence and in noise in humans is difficult, if not impossible, to date with the conventional methods available. That is why in certain situations, the hearing aids of patient with hearing loss fail, especially in the presence of noise.

In this study the investigators aim at investigating the global spontaneous and sound evoked human auditory nerve activity from electrophysiological acquisitions performed directly on the cochlear nerve in patients requiring posterior fossa surgery.

DETAILED DESCRIPTION:
The fine evaluation of the function of auditory neurons in silence and in noise in humans is difficult, if not impossible, to date with the conventional methods available. That is why in certain situations, the hearing aids of patient with hearing loss fail, especially in the presence of noise.

In this study the investigators aim at investigating the global spontaneous and sound evoked human auditory nerve activity from electrophysiological acquisitions performed directly on the cochlear nerve in patients requiring posterior fossa surgery.

Stimulations will be performed in silence and in noise from stimuli identical to those used during the preoperative auditory assessment: clic and speech syllable stimulation. These acquisitions will allow us to compare clinical and electrophysiological data in order to better understand the coding of hearing in normal and hearing loss humans under silent and noisy conditions. A prospective longitudinal study will be performed.

ELIGIBILITY:
inclusion criteria :

Will be included as hearing impaired patients:

* male or female
* over 18 years of age
* who are to undergo surgery on the cerebellopontine angle (microvascular decompression, vestibular neurotomy, removal of a meningioma or schwannoma tumor)
* with a mild to severe sensorineural hearing loss defined by an average hearing loss (average of thresholds obtained at 500, 1000, 2000 and 4000 Hz) greater than 20 dB and less than 90 dB in pure tone bone conduction audiometry on the side of the operated ear.
* affiliated to a social security system.
* have read the information note describing the study and have agreed in writing to participate by signing the informed consent form.

Will be included as normal hearing patients:

* male or female
* over 18 years of age
* who are to undergo surgery in the cerebellopontine angle (microvascular decompression, vestibular neurotomy, removal of a meningioma or schwannoma tumor)
* free of neuro-sensory deafness, defined by average hearing thresholds less than or equal to 20 dB in tonal bone conduction audiometry on the side of the operated ear
* affiliated with a social security system.
* having read the information note describing the study and having agreed in writing to participate by signing the informed consent form.

exclusion criteria :

Patients for whom the auditory nerve is not accessible during surgery,

* because of a complete tumor invasion of the cochlear nerve (stage III and IV neuroma, advanced meningioma)
* because of an anatomical feature not identified during the preoperative examination, making its exposure for recordings impossible (protrusion of the posterior face of the rock)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2027-06-07 (Estimated); Study Completion 2027-06-07 (Estimated)

PRIMARY OUTCOMES:
Compare the amplitude of global evoked auditory nerve activity | 66 months
  Compare the amplitude and spectrum of global evoked auditory nerve activity in silence and in noise with basic and speech stimuli between patients defined as normo and hearing loss based on preoperative audiometric tests.
Compare the spectrum of global evoked auditory nerve activity | 66 months
  Compare the spectrum of global evoked auditory nerve activity in silence and in noise with basic and speech stimuli between patients defined as normo and hearing loss based on preoperative audiometric tests

SECONDARY OUTCOMES:
Compare the difference of coding of the temporal envelope | 66 months
  Compare the difference of coding of the temporal envelope of the collected signal in the normo and hearing impaired groups.
Compare the difference of coding of the fine structure | 66 months
  Compare the difference of coding of the fine structure of the collected signal in the normo and hearing impaired groups.
Compare the two groups of investigation | 66 months
  To investigate within the group of normo hearing patients whether the amplitude of global evoked auditory nerve activity is different between those with the best and worst results in the pre-operative vocal speech in noise test.
Compare the two groups of investigation | 66 months
  To investigate within the group of normo hearing patients whether the spectrum of global evoked auditory nerve activity is different between those with the best and worst results in the pre-operative vocal speech in noise test.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France